CLINICAL TRIAL: NCT02080299
Title: Protection of Heart, Brain and Kidney by Remote Ischemic Preconditioning in Patients Undergoing Transcatheter Aortic Valve Implantation - a Randomized, Single-blind Study
Brief Title: Protection by Remote Ischemic Preconditioning During Transcatheter Aortic Valve Implantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Essen (Other)
Collaborators: Koblenz University of Applied Science (Other)
Responsible Party: Principal Investigator, Philipp Kahlert, MD, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 135355-BO
Record Dates: First submitted 2014-03-01; First posted 2014-03-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemic preconditioning (RIPC) (Active Comparator): RIPC-protocol before TAVI: after induction of conscious sedation/anesthesia, but prior to TAVI procedure, remote ischemic preconditioning (RIPC) protocol is performed, consisting of 3 cycles of 5 minutes left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 minutes of reperfusion, followed by a time interval between the end of the last deflation and local groin anaesthesia with subsequent skin puncture of 30 min.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- Placebo (Placebo Comparator): Placebo protocol before TAVI: After induction of conscious sedation/anesthesia and before TAVI, the cuff is left uninflated for 30 min, followed by a further time interval of 30 min until local groin anaesthesia with subsequent skin puncture.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — 3 circles of 5 min left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 min reperfusion, preceding TAVI procedure.
  Arms: Remote ischemic preconditioning (RIPC)
Procedure: Placebo — Prior to TAVI-procedure, the blood pressure cuff remains uninflated for 30 min.
  Arms: Placebo

SUMMARY:
Transcatheter aortic valve implantation (TAVI) has rapidly been adopted into clinical practice, but concerns have been raised regarding periprocedural complications like e.g. myocardial injury, stroke or acute kidney injury. Remote ischemic preconditioning (RIPC) with upper limb ischemia/reperfusion provides perioperative myocardial protection in patients undergoing elective coronary artery bypass surgery. The present study assesses protection of heart, brain and kidney by RIPC in patients undergoing TAVI. The study also addresses safety and clinical outcome.

DETAILED DESCRIPTION:
* On the assumption of our recent data (Thielmann et al, Lancet 2013, 382(9892):597-604), we performed a power analysis, revealing an estimated enrollment of 189 patients per group. But since no true data exist regarding RIPC and TAVI, interim analysis will be performed after 50 patients per group.
* After induction of conscious sedation or general anaesthesia, RIPC is accomplished by 3 cycles of 5 min inflation/5 min deflation of a blood pressure cuff around the left arm to 200 mm Hg. In the placebo group, the blood pressure cuff remains uninflated for 30 min.
* Blind: study coordinators, outcome assessors, operators and treating physicians except for the attending anaesthetist.
* Drugs used for conscious sedation: midazolam, remifentanil.
* Drugs used for general anaesthesia: sufentanil, etomidate, rocuronium, isoflurane.
* TAVI is performed by standard techniques using the balloon-expandable Sapien XT (Edwards Lifesciences Inc., Irvine, California, USA) and the next-generation Sapien 3 stent-valve bioprosthesis which replaces the Sapien XT prosthesis, when CE-approved.
* Arterial blood samples are obtained prior to and after RIPC-maneuver/Placebo, after aortic valve implantation and after access site closure, for biochemical analyses focussing on ligands that have been previously implicated in conditioning protocols at various organs. A bioassay system, consisting of a Langendorff-perfused isolated heart with ischemia and reperfusion will be used. This bioassay system will be exposed to the obtained arterial plasma of the patients.
* Venous blood samples are drawn before TAVI and at 1, 6, 12, 24, 48 and 72 hours after the procedure.
* Cardiac and cerebral MRI is performed in selected patients at baseline and within the first week after TAVI.
* On-site follow-up at 3±3 months, 12±3 months and yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with severe symptomatic native aortic valve stenosis scheduled for elective TAVI due to a prohibitive or high risk for surgical aortic valve replacement as judged by the institutional heart team based on risk scores and comorbidity assessment
* Written informed consent

Exclusion Criteria:

* Life expectancy < 1 year
* Patients who are unlikely to gain improvement in their quality of life by TAVI procedure
* Unfavorable anatomy for TAVI (e.g. inadequate annulus size)
* Left-ventricular thrombus
* Active endocarditis
* Active infection
* Acute ST-segment elevation myocardial infarction
* Hemodynamic instability
* Preoperative troponin I concentration above the upper normal limit of 0.1 ng/ml
* Stroke within the last 6 weeks
* Acute or chronic hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Extent of periinterventional myocardial injury as reflected by the geometric mean of the area under the curve (AUC) for troponin I serum concentrations | 72 hours postinterventionally after TAVI

SECONDARY OUTCOMES:
Periprocedural myocardial infarction according to current Valve Academic Research Consortium (VARC-2) criteria | 72 hours postinterventionally after TAVI
Incidence of new wall abnormalities and deterioration of overall left ventricular function as assessed by postinterventional transthoracic echocardiography | Within the first week after TAVI
Incidence of new-onset cardiac arrhythmias including the necessity of defibrillation or transient/permanent pacemaker implantation as assessed by continuous ECG-monitoring | Within the first week after TAVI
Prevalence and volume of delayed gadolinium enhancement | Within the first week after TAVI
  Cardiac MRI will be performed in selected patients.
Maximum elevation of serum creatinine concentration | Until 72 hours after TAVI
Maximum decrease of estimated glomerular filtration rate | Until 72 hours after TAVI
Incidence of VARC-2 defined acute kidney injury | Until 72 hours after TAVI and until discharge
Total and median per patient number as well as total and median per patient volume of new foci of restricted diffusion | Within the first week after TAVI
  Cerebral MRI will be performed in selected patients.
Cardioprotective factor release into circulating blood | Day of intervention
  Blood samples will be collected at 4 time points: prior to and after RIPC-maneuver/Placebo, after aortic valve implantation and after access site closure. Time frame: approximately 2,5 hours.
All cause mortality and major adverse cardiac and cerebrovascular events (MACCE) at 30 days | Within the first 30 days after TAVI
All cause mortality and major adverse cardiac and cerebrovascular events (MACCE) at 1 year | Within the first year after TAVI
All cause mortality and major adverse cardiac and cerebrovascular events (MACCE) after 3 months | Until 3 months after TAVI
VARC-2 defined combined early TAVI safety endpoint at 30 days | Until 30 days after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kahlert, MD, Principal Investigator — Department of Cardiology, West-German Heart Center Essen, University Duisburg-Essen; Matthias Thielmann, MD, Principal Investigator — Department of Thoracic and Cardiovascular Surgery, West-German Heart Center Essen, University Duisburg-Essen; Petra Kleinbongard, PhD, Principal Investigator — Institute of Pathophysiology, University Duisburg-Essen; Eva Kottenberg, MD, Principal Investigator — Clinic for Anesthesiology and Intensive Care Medicine, University Duisburg-Essen; Jürgen Peters, MD, Principal Investigator — Clinic for Anesthesiology and Intensive Care Medicine, University Duisburg-Essen; Heinz Jakob, MD, Principal Investigator — Department of Thoracic and Cardiovascular Surgery, West-German Heart Center Essen, University Duisburg-Essen; Raimund Erbel, MD, Principal Investigator — Department of Cardiology, West-German Heart Center Essen, University Duisburg-Essen; Gerd Heusch, MD, PhD, Principal Investigator — Institute of Pathophysiology, University Duisburg-Essen
Locations (1):
- Department of Cardiology, West-German Heart Center Essen, University Duisburg-Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thielmann M, Kottenberg E, Boengler K, Raffelsieper C, Neuhaeuser M, Peters J, Jakob H, Heusch G. Remote ischemic preconditioning reduces myocardial injury after coronary artery bypass surgery with crystalloid cardioplegic arrest. Basic Res Cardiol. 2010 Sep;105(5):657-64. doi: 10.1007/s00395-010-0104-5. Epub 2010 May 21. PMID 20495811
- [Background] Kottenberg E, Thielmann M, Bergmann L, Heine T, Jakob H, Heusch G, Peters J. Protection by remote ischemic preconditioning during coronary artery bypass graft surgery with isoflurane but not propofol - a clinical trial. Acta Anaesthesiol Scand. 2012 Jan;56(1):30-8. doi: 10.1111/j.1399-6576.2011.02585.x. Epub 2011 Nov 21. PMID 22103808
- [Background] Heusch G, Musiolik J, Kottenberg E, Peters J, Jakob H, Thielmann M. STAT5 activation and cardioprotection by remote ischemic preconditioning in humans: short communication. Circ Res. 2012 Jan 6;110(1):111-5. doi: 10.1161/CIRCRESAHA.111.259556. Epub 2011 Nov 23. PMID 22116817
- [Background] Kottenberg E, Musiolik J, Thielmann M, Jakob H, Peters J, Heusch G. Interference of propofol with signal transducer and activator of transcription 5 activation and cardioprotection by remote ischemic preconditioning during coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2014 Jan;147(1):376-82. doi: 10.1016/j.jtcvs.2013.01.005. Epub 2013 Mar 1. PMID 23465551
- [Background] Thielmann M, Kottenberg E, Kleinbongard P, Wendt D, Gedik N, Pasa S, Price V, Tsagakis K, Neuhauser M, Peters J, Jakob H, Heusch G. Cardioprotective and prognostic effects of remote ischaemic preconditioning in patients undergoing coronary artery bypass surgery: a single-centre randomised, double-blind, controlled trial. Lancet. 2013 Aug 17;382(9892):597-604. doi: 10.1016/S0140-6736(13)61450-6. PMID 23953384
- [Background] Kleinbongard P, Thielmann M, Jakob H, Peters J, Heusch G, Kottenberg E. Nitroglycerin does not interfere with protection by remote ischemic preconditioning in patients with surgical coronary revascularization under isoflurane anesthesia. Cardiovasc Drugs Ther. 2013 Aug;27(4):359-61. doi: 10.1007/s10557-013-6451-3. No abstract available. PMID 23440355
- [Background] Kahlert P, Knipp SC, Schlamann M, Thielmann M, Al-Rashid F, Weber M, Johansson U, Wendt D, Jakob HG, Forsting M, Sack S, Erbel R, Eggebrecht H. Silent and apparent cerebral ischemia after percutaneous transfemoral aortic valve implantation: a diffusion-weighted magnetic resonance imaging study. Circulation. 2010 Feb 23;121(7):870-8. doi: 10.1161/CIRCULATIONAHA.109.855866. PMID 20177005
- [Derived] Kahlert P, Hildebrandt HA, Patsalis PC, Al-Rashid F, Janosi RA, Nensa F, Schlosser TW, Schlamann M, Wendt D, Thielmann M, Kottenberg E, Frey U, Neuhauser M, Forsting M, Jakob HG, Rassaf T, Peters J, Heusch G, Kleinbongard P. No protection of heart, kidneys and brain by remote ischemic preconditioning before transfemoral transcatheter aortic valve implantation: Interim-analysis of a randomized single-blinded, placebo-controlled, single-center trial. Int J Cardiol. 2017 Mar 15;231:248-254. doi: 10.1016/j.ijcard.2016.12.005. Epub 2016 Dec 6. PMID 27940009